CLINICAL TRIAL: NCT06648057
Title: Investigation of Predictive Biomarkers in Patients With Advanced Biliary Tract Cancer Treated With Lenvatinib Plus Pembrolizumab
Brief Title: Investigation of Predictive Biomarkers in Patients With Advanced BTC Treated With Lenvatinib Plus Pembrolizumab
Status: Recruiting | Type: Observational
Sponsor: CHA University (Other)
Responsible Party: Principal Investigator, Hong Jae Chon, Principal Investigator, CHA University
Other Study IDs: CHAMC 2024-08-040
Record Dates: First submitted 2024-10-07; First posted 2024-10-18 (Actual); Last update posted 2024-10-18 (Actual); Status verified 2024-10

CONDITIONS: Biliary Tract Cancer; Cholangiocarcinoma
Keywords: Lenvatinib; Pembrolizumab; Biliary Tract Cancer; Biomarker; RNA sequencing
MeSH Terms: conditions — Biliary Tract Neoplasms; Cholangiocarcinoma | interventions — lenvatinib; pembrolizumab; Liquid Biopsy; Base Sequence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tissue, Blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Len/Pemb: lenvatinib plus pembrolizumab combination therapy.
  Interventions: Drug: lenvatinib plus pembrolizumab

INTERVENTIONS:
Drug: lenvatinib plus pembrolizumab — * The collection of peripheral blood samples will follow the schedule below (20 cc per collection, up to 5 times):
  * Before systemic therapy, at 3 weeks after starting systemic therapy (Cycle 1), at 6 weeks (Cycle 2)
  * (If possible) at the time of confirmed partial response (1 time), and at the time of disease progression (1 time).
  * Additional tumor tissue samples will be collected only if possible, according to the following schedule:
  If the patient undergoes surgery or additional biopsy related to treatment (collected from preserved specimens).
  Other Names: Liquid biopsy, RNA-sequencing, NGS

SUMMARY:
The goal of this observational study is to evaluate the clinical efficacy and safety of lenvatinib plus pembrolizumab combination therapy in patients with advanced biliary tract cancer (BTC). This study aims to identify potential biomarkers that may predict treatment response by analyzing genetic data from blood and tissue samples. The study will focus on real-world clinical outcomes and the exploratory discovery of biomarkers associated with the efficacy of this treatment regimen.

DETAILED DESCRIPTION:
Biliary tract cancers (BTCs) have a higher prevalence in Asia compared to Western countries, with South Korea ranking second globally in BTC incidence. According to data from the Central Cancer Registry in 2023, the 5-year survival rate for BTC from 2017 to 2021 was 28.9%, significantly lower than other cancers such as gastric cancer (77.9%), colorectal cancer (74.3%), and breast cancer (93.8%).

Surgery is the primary treatment for BTC, but only 40-50% of patients are eligible for curative resection. For patients with unresectable, advanced, or metastatic BTC, the standard first-line treatment has been gemcitabine plus cisplatin (GP) since the results of the ABC-02 Phase 3 trial in 2010. Recently, two Phase 3 trials-TOPAZ-1 in 2022 and KEYNOTE-966 in 2023-demonstrated significant survival benefits with the addition of immune checkpoint inhibitors (durvalumab or pembrolizumab) to GP therapy, establishing these combination regimens as the new first-line standard treatment for advanced BTC. These combinations have been approved for use in South Korea.

However, for patients who fail first-line GP therapy, the most commonly selected second-line treatment, FOLFOX (5-FU + leucovorin + oxaliplatin), offers only a modest survival extension of about one month compared to supportive care. This highlights the clinical unmet need for more effective second-line treatments. A multicenter Phase 2 trial has demonstrated the efficacy of lenvatinib plus pembrolizumab as a promising treatment option for these patients.

This prospective observational study aims to evaluate the clinical efficacy and safety of lenvatinib plus pembrolizumab combination therapy in real-world clinical practice for advanced BTC. Additionally, the study seeks to explore potential predictive biomarkers through genetic analyses of blood and tissue samples to better understand which patients are most likely to benefit from this treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically or cytologically confirmed advanced biliary tract cancer.
* Patients scheduled to receive Lenvatinib + Pembrolizumab for the treatment of advanced biliary tract cancer.
* ECOG performance status of 0-2.
* Patients aged 20 years or older at the time of treatment initiation.
* Patients who understand and consent to participate in this study, and agree to provide samples obtained during the examination process.

Exclusion Criteria:

* Patients who do not consent to participate in the study or withdraw their consent.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Advenced Biliary Tract Cancer will be recruited at CHA Bundang Medical Center
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-09-23 (Actual); Primary Completion 2026-09-23 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
collected tumor samples | through study competition, an average of 2 years
  Tumor samples will be collected from patients with advanced biliary tract cancer. The incidence of genetic alterations in these samples will be analyzed using H&E staining, immunohistochemistry (IHC), and RNA sequencing. The data will be reported as the percentage of patients with detectable genetic alterations and correlated with treatment response and survival duration.
Collected Blood Samples | Through study completion, an average of 2 years
  Blood samples will be collected from patients with advanced biliary tract cancer.These samples will undergo flow cytometry, ELISA, and ctDNA analysis, and the results will be correlated with treatment response and survival outcomes. (PFS, OS).

SECONDARY OUTCOMES:
Multi-Omics Analysis for Therapeutic Target Identification | Through study completion, an average of 2 years.
  Multi-omics analysis, including DNA, RNA, and protein analysis, will be conducted to identify potential therapeutic targets and subtypes of biliary tract cancer. The analysis will integrate molecular data to identify actionable genetic alterations and protein expression levels, which will be summarized and correlated with clinical outcomes (e.g., PFS, OS).
Biomarkers on the Efficacy of Lenvatinib and Pembrolizumab for Advanced Biliary Tract Cancer | Through study completion, an average of 2 years.
  his outcome will investigate the correlation between molecular biomarkers and the efficacy of lenvatinib and pembrolizumab in patients with advanced biliary tract cancer. Biomarkers will be evaluated for their association with overall survival (OS), progression-free survival (PFS), and objective response rate (ORR). The outcome will report which biomarkers predict better therapeutic response.

OTHER OUTCOMES:
Progression-Free Survival (PFS) | Through study completion, an average of 2 years.
  This outcome measures the time from the start of treatment to the first occurrence of disease progression or death. PFS will be analyzed using Kaplan-Meier survival curves, and the median PFS will be reported.
Overall Survival (OS) | Through study completion, an average of 2 years.
  This outcome measures the time from the start of treatment to death from any cause. OS will be evaluated and reported using Kaplan-Meier survival analysis, and median OS will be calculated.
Objective Response Rate (ORR) | Through study completion, an average of 2 years.
  ORR is defined as the percentage of patients who achieve a complete or partial response based on RECIST 1.1 criteria. This outcome will report the proportion of patients who show a measurable response to treatment.
Incidence of Adverse Events (AEs) | Through study completion, an average of 2 years.
  The safety and tolerability of lenvatinib and pembrolizumab will be assessed by monitoring the occurrence and severity of adverse events, graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Hong Jae Chon, MD. PhD, Principal Investigator — CHA University
Locations (1):
- Bundang CHA Medical Center, Seongnam-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Valle J, Wasan H, Palmer DH, Cunningham D, Anthoney A, Maraveyas A, Madhusudan S, Iveson T, Hughes S, Pereira SP, Roughton M, Bridgewater J; ABC-02 Trial Investigators. Cisplatin plus gemcitabine versus gemcitabine for biliary tract cancer. N Engl J Med. 2010 Apr 8;362(14):1273-81. doi: 10.1056/NEJMoa0908721. PMID 20375404
- [Result] Oh DY, Ruth He A, Qin S, Chen LT, Okusaka T, Vogel A, Kim JW, Suksombooncharoen T, Ah Lee M, Kitano M, Burris H, Bouattour M, Tanasanvimon S, McNamara MG, Zaucha R, Avallone A, Tan B, Cundom J, Lee CK, Takahashi H, Ikeda M, Chen JS, Wang J, Makowsky M, Rokutanda N, He P, Kurland JF, Cohen G, Valle JW. Durvalumab plus Gemcitabine and Cisplatin in Advanced Biliary Tract Cancer. NEJM Evid. 2022 Aug;1(8):EVIDoa2200015. doi: 10.1056/EVIDoa2200015. Epub 2022 Jun 1. PMID 38319896
- [Result] Kelley RK, Ueno M, Yoo C, Finn RS, Furuse J, Ren Z, Yau T, Klumpen HJ, Chan SL, Ozaka M, Verslype C, Bouattour M, Park JO, Barajas O, Pelzer U, Valle JW, Yu L, Malhotra U, Siegel AB, Edeline J, Vogel A; KEYNOTE-966 Investigators. Pembrolizumab in combination with gemcitabine and cisplatin compared with gemcitabine and cisplatin alone for patients with advanced biliary tract cancer (KEYNOTE-966): a randomised, double-blind, placebo-controlled, phase 3 trial. Lancet. 2023 Jun 3;401(10391):1853-1865. doi: 10.1016/S0140-6736(23)00727-4. Epub 2023 Apr 16. PMID 37075781
- [Result] Lamarca A, Palmer DH, Wasan HS, Ross PJ, Ma YT, Arora A, Falk S, Gillmore R, Wadsley J, Patel K, Anthoney A, Maraveyas A, Iveson T, Waters JS, Hobbs C, Barber S, Ryder WD, Ramage J, Davies LM, Bridgewater JA, Valle JW; Advanced Biliary Cancer Working Group. Second-line FOLFOX chemotherapy versus active symptom control for advanced biliary tract cancer (ABC-06): a phase 3, open-label, randomised, controlled trial. Lancet Oncol. 2021 May;22(5):690-701. doi: 10.1016/S1470-2045(21)00027-9. Epub 2021 Mar 30. PMID 33798493
- [Result] Shi C, Li Y, Yang C, Qiao L, Tang L, Zheng Y, Chen X, Qian Y, Yang J, Wu D, Xie F. Lenvatinib Plus Programmed Cell Death Protein-1 Inhibitor Beyond First-Line Systemic Therapy in Refractory Advanced Biliary Tract Cancer: A Real-World Retrospective Study in China. Front Immunol. 2022 Jul 27;13:946861. doi: 10.3389/fimmu.2022.946861. eCollection 2022. PMID 35967452
- [Result] Lin J, Yang X, Long J, Zhao S, Mao J, Wang D, Bai Y, Bian J, Zhang L, Yang X, Wang A, Xie F, Shi W, Yang H, Pan J, Hu K, Guan M, Zhao L, Huo L, Mao Y, Sang X, Wang K, Zhao H. Pembrolizumab combined with lenvatinib as non-first-line therapy in patients with refractory biliary tract carcinoma. Hepatobiliary Surg Nutr. 2020 Aug;9(4):414-424. doi: 10.21037/hbsn-20-338. PMID 32832493
- [Result] Li L, Yu D, Yang J, Zhang F, Zhang D, Lin Z, Zhai M, Wang J, Zhang T, Zhao L. Significant response to pembrolizumab plus lenvatinib in Epstein-Barr-virus-associated intrahepatic cholangiocarcinoma: a case report. Cancer Biol Ther. 2024 Dec 31;25(1):2338644. doi: 10.1080/15384047.2024.2338644. Epub 2024 Apr 22. PMID 38650446